CLINICAL TRIAL: NCT06274632
Title: ADELANTE: A Randomized Controlled Trial of an Intervention to Improve Engagement in Care for Latinos With HIV
Brief Title: ADELANTE: A Randomized Controlled Trial to Improve Engagement in Care for Latinos With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Baylor College of Medicine (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Julie H Levison, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023P001913
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS
Keywords: Latino; Hispanic; HIV/AIDS; health outcomes; community health worker
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADELANTE (Experimental): Participants will receive 5, individualized problem solving sessions delivered by a community health worker over 6 months. The intervention content is framed around a bi-lingual film about HIV.
  Interventions: Behavioral: ADELANTE
- Enhanced Care Condition (No Intervention): Participants in the enhanced care control group will receive 5 locator phone calls confirming contact information at the same interval as CHW sessions in the ADELANTE group. They will be offered routine HIV health promotion materials as is available in the clinic. If a participant requests support for navigation or case management, they will be encouraged to contact their HIV team

INTERVENTIONS:
Behavioral: ADELANTE — A manualized problem-solving intervention that addresses barriers to viral suppression in Latinos with HIV. At the patient-level, CHWs use motivational interviewing to facilitate problem-solving skill development around attending HIV care and adherence and establish an individually tailored goal-setting plan. We target emotional well-being and self-management through a rapport with CHW and the integration of an HIV-centered telenovela to facilitate participant reflection on difficult topics for skill-building. The CHW will also link the participant to needed services.
  Arms: ADELANTE

SUMMARY:
The goal of this study is to test the effectiveness of ADELANTE on viral suppression among Latinos with HIV and viral non-suppression. Participants will receive ADELANTE (5-session, community health worker-delivered, problem-solving intervention) or enhanced care condition (ECC, 5 reminder phone calls). We will evaluate the overall effectiveness of ADELANTE compared with ECC on rates of viral suppression and emergency room visits and hospitalizations. Our hypothesis is that ADELANTE participants will achieve higher rates of viral suppression and will have lower rates of emergency room visits and hospitalizations compared with ECC at 12 months post-randomization.

DETAILED DESCRIPTION:
Participants will be Latinx/Hispanic individuals age ≥18 years who are at least 3 months since initiation of HIV treatment and have evidence of viral non-suppression (HIV RNA ≥200 cpm). Participants will be recruited from two Ryan White-funded clinics in geographic priority areas in the US Ending the HIV Epidemic (EHE) Plan due to high HIV incidences and prevalence. In the intervention, a bilingual (English-Spanish speaking) community health worker (CHW) will deliver a manualized problem-solving intervention that is framed around an HIV-focused telenovela, or drama-based film. The CHW will deliver five sessions within 6 months. The CHW will assist in problem-solving to improve behavioral activation and self-management skills and help participants adhere to HIV treatment and attend medical appointments. The CHW will also link patients to resources. In the enhanced care condition, participants will receive 5 phone calls. They will not receive the intervention or access to navigation beyond routine care. Measurements will occur at baseline, month-3, month-6, and month-12 post randomization by study staff blinded to the allocation status of participants. Participants will be remunerated for each assessment.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latino/Latina/Latinx/Hispanic; adults 18 years and over; with HIV infection confirmed by standard laboratory results available in the medical record; 3 or more months from initial entry into care with a medical provider who can prescribe HIV antiretroviral treatment; receiving HIV primary care at Jackson Memorial Hospital or Thomas Street at Quentin Mease Health Center/Harris Health System; and medical record evidence with last viral load (VL) indicating viral non-suppression (HIV RNA ≥200 cpm) within 12 months prior to assessment of eligibility, as it is typical for providers to obtain laboratories prior to a clinic visit in preparation for counseling.

Exclusion Criteria:

* Lacks capacity to consent (measured by a validated screener), plans to move out of the county in the next 6 months, or currently participating in an HIV intervention study with ongoing follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
12-month viral suppression | month-12
  Viral suppression is defined as number of participants with HIV RNA less than 200 cpm. Response determined by viral load values in the medical record closest to the scheduled 12-month date, allowing for a range of three months before or after the scheduled 12-month date.

SECONDARY OUTCOMES:
Number of Emergency department visits | 12 months
  All-cause emergency department visits
Number of Hospitalizations | 12 months
  All-cause hospitalizations defined as number of different times stayed in any hospital overnight or longer
6-month viral suppression | month-6
  Viral suppression is defined as number of participants with HIV RNA less than 200 cpm. Response determined by viral load values in the medical record closest to the scheduled 6-month date, allowing for a range between 4 and 8 months.
Retention in care | 12 months
  A dichotomized outcome (yes/no) with yes defined as at least one visit to the clinic providing HIV treatment at both time periods (months 0-6 and months 7-12) with the two visits at least 90 days apart and no defined as no HIV visit from at least one time period. Attendance determined by review of the medical record.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Baylor College of Medicine, Houston, Texas